CLINICAL TRIAL: NCT01848977
Title: Comparison of Two Devices Using Near-infra Red Spectroscopy for the Measurement of Tissue Oxygenation During a Vascular Occlusion Test (INVOS® Versus Inspectra™)
Brief Title: Comparison of Two Devices Using Near-infra Red Spectroscopy During a Vascular Occlusion Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Ph.D., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: H-1302-016-462
Record Dates: First submitted 2013-04-07; First posted 2013-05-08 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Measures; near-Infrared spectroscopy; ischemia; reperfusion
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- vascular occlusion test (Experimental): The pediatric SomaSensor™ probe of INVOS® and the 15-mm sensor of InSpectra™ are placed on each thenar muscle in the same subject. The side on which the probe will be placed is randomly determined. INVOS® updates data every 5 s and data (SrO2) will be manually recorded. The data of InSpectra™ (StO2) are automatically collected and sampled every 2 s.
  Vascular occlusion test (VOT) is done as follows:Adult-size blood pressure cuffs are placed around each upper arm. The both cuffs are simultaneously inflated to 30 mmHg above the initial systolic blood pressure and kept inflated until the SrO2 or StO2 decreased to 40%. When the value reaches 40% or just below it, the cuff on the same side is deflated rapidly. The data will be collected until the SrO2 and StO2 values returned to the baseline.
  Interventions: Device: vascular occlusion test

INTERVENTIONS:
Device: vascular occlusion test — Using Invos® probe attacted to one thenar muscle, tissue oxgyenation is measured by VOT.
Device: vascular occlusion test — Using Inspectra™ probe attacted to another thenar muscle, tissue oxgyenation is measured by VOT.

SUMMARY:
Tissue oxygen saturation is non-invasively measured using near-infrared spectroscopy, by two device, INVOS®(somanetics Corporation, USA ) and InSpectra™ (Hutchinson Technology, USA). Each probes are attached to both thenar muscles and vascular occlusion test (VOT) is performed. The investigators will compare the Invos® data to InSpectra™ to investigate whether tissue oxygen saturation values by INVOS® can substitute for InSpectra™.

DETAILED DESCRIPTION:
Tissue oxygen saturation is non-invasively measured using near-infrared spectroscopy, by two device, INVOS®(somanetics Corporation, USA ) and InSpectra™ (Hutchinson Technology, USA). InSpectra™ was introduced later than INVOS®.

With InSpectra™, clinicians have used a vascular occlusion test (VOT) to evaluate dynamic changes in tissue oxygen saturation during ischemia and reperfusion, and thus, microcirculatory function. There have been little data about VOT using INVOS®, although it is more popular device.

We hypothesized that there would be a difference between the values from INVOS® and InSpectra™. The aim of this study is to evaluate changes in tissue oxygen saturation in the thenar muscle during VOT using INVOS® and comapre it to InSpectra™ in a normal population.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject

Exclusion Criteria:

* age under 18 years old
* with arteriovenous fistula
* with peripheral vessel disease
* taking vasoactive drug
* with a skin ailment
* with HTN, DM
* with diagnosed heart disease

Ages: 26 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Ph.D., Study Director — Seoul National University Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vascular Occlusion Test
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vascular Occlusion Test
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Change of Tissue Oxygenation Value During Ischemia and Reperfusion Period Until Basline Value Was Achieved
Description: During vascular occlusion test, the changes of StO2 and SrO2 values can divided into 3 epoch; Desaturation, Reoxygenation and Reactive hyperemia. After data collection, the rate of desaturation and reoxygenation were calculated.
Time Frame: Until basline tissue oxygenation value was achieved
Measure: Mean (Standard Deviation); unit: %/min
Groups:
- INVOS®: Data from INVOS® during VOT were manually recorded. Desaturation and reoxygenation rate were calculated and compared to InSpectra™ .
- InSpectra™: Data from InSpectra™ during VOT were manually recorded. Desaturation and reoxygenation rate were calculated and compared to INVOS®.
Arm/Group | INVOS® | InSpectra™
Number analyzed (Participants) | 20 | 20
%/min
  Desaturation rate | 17.9 (2.3) | 13.5 (2.1)
  Reoxygenation rate | 280.0 (57.5) | 186.5 (39.7)
Statistical Analysis 1: Comparison: INVOS® vs InSpectra™; Unpaired t-test was used to compare the difference between SrO2 and StO2; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Baseline, Miminum and Maximum Tissue Oxygenation Value Measured by INVOS® (SrO2) Until Basline Value Was Achieved
Description: Before VOT. basline StO2 and SrO2 were recorded and compared each other. During VOT, minimum/maximum StO2 and SrO2 were also recorded and compared each other.
Time Frame: Until basline tissue oxygenation value was achieved
Measure: Mean (Standard Deviation); unit: percentage of oxyhemoglobin
Groups:
- INVOS®: Basline value before VOT,and minimum/ maximum values of INVOS® were obtained and compared to InSpectra™ .
- InSpectra™: Basline value before VOT,and minimum/ maximum values of InSpectra™ were obtained and compared to INVOS®.
Arm/Group | INVOS® | InSpectra™
Number analyzed (Participants) | 20 | 20
percentage of oxyhemoglobin
  baseline value before VOT | 75.6 (8.2) | 81.8 (3.4)
  minimum value during VOT | 39.6 (0.5) | 40.2 (0.4)
  maximum value during VOT | 95.1 (0.2) | 94.6 (1.7)

3. Primary Outcome: Sum of Tissue Oxygenation Value Which Above Basline Value After Reperfusion Period Until Basline Value Was Achieved
Description: as for outcome 1
Time Frame: Until basline tissue oxygenation value was achieved
Measure: Mean (Standard Deviation); unit: %*min
Groups:
- INVOS®: Data from INVOS® during VOT were manually recorded. Reactive hyperemic area were calculated and compared to InSpectra™ .
- InSpectra™: Data from InSpectra™ during VOT were manually recorded. Reactive hyperemic area were calculated and compared to INVOS®.
Arm/Group | INVOS® | InSpectra™
Number analyzed (Participants) | 20 | 20
%*min | 23.5 (9.6) | 16.4 (6.3)

ADVERSE EVENTS:
Time Frame: up to 1 days after study
Arm/Group | Vascular Occlusion Test
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No